CLINICAL TRIAL: NCT05095506
Title: Initial Evaluation of an eHealth Self-Management System to Reduce Depression and Increase Resilience After SCI (SCIRP Pilot Clinical Trial)
Brief Title: Evaluation of an eHealth System to Reduce Depression and Increase Resilience After SCI
Acronym: SCIRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Kessler Foundation (Other); Department of Veterans Affairs, New Jersey (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Tulsky, Professor and Director, Center for Health Assessment Research and Translation, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1564112; W81XWH-20-1-0786 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2021-10-22; First posted 2021-10-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHeatlh Intervention Arm (Experimental): The intervention platform is an interactive, web-based self-management program comprised of computer-adaptive tests (CATs) to assess depression, anxiety, and resilience and multimedia-assisted components. Participants will access the system once a week for 6 weeks, complete the symptom monitoring CATs, receive score reports, and watch a system-assigned self-management strategy video (which is selected by the system based on the participant's current level of depression/anxiety symptoms).
  Interventions: Other: eHealth Intervention
- Active Control Arm (Active Comparator): The active control condition is a static web-based program which also includes computer-adaptive tests (CATs) to assess depression, anxiety, and resilience, but does not provide score reports and plays a predetermined educational video (related to health promotion after SCI) each week. Participants will access the system once a week for 6 weeks, complete the symptom monitoring CATs and watch the educational video.
  Interventions: Other: Active Control Condition

INTERVENTIONS:
Other: eHealth Intervention — The intervention platform is interactive, and uses multimedia-assisted components. The system uses three SCI-QOL computer-adaptive tests (CATs) to assess depression, anxiety, and resilience; cut scores are used to tailor multi-media content that specifically addresses users' emotional health concerns.
  Arms: eHeatlh Intervention Arm
Other: Active Control Condition — The active control condition is a static site that displays symptom assessments followed by one educational video each week. These videos, which play in a predetermined order, provide education about managing physical health in individuals with SCI.
  Arms: Active Control Arm

SUMMARY:
The availability of symptom monitoring and self-management (SMSM) interventions is especially important for civilians and military populations with spinal cord injuries (SCI). High rates of depressive disorders (20-40%) and anxiety disorders (20-25%) have been found in both civilian and military populations and are significant contributors to both quality of life and well-being after SCI. Previous self-management interventions targeting physical activity and self-reliance in individuals with SCI have demonstrated significant health and lifestyle benefits. However, it has been shown that the injured individual's psychological outlook and mood can either enable or hinder self-management efforts and that currently available SCI-specific self-management programs may be inadequate. Developing interventions to reduce mental health symptoms following SCI is therefore critical to improve the lives of individuals, alleviate resource strain on military and civilian health care systems, and potentially reduce the rate of mortality by suicide in Veterans and civilians living with SCI. The current study will build on prior work developing an intervention platform to assess the effectiveness of this eHealth SMSM system and will test the feasibility and effectiveness of the intervention platform.

ELIGIBILITY:
Inclusion Criteria:

* Access to the internet and an internet-enabled device
* Diagnosis of a sudden-onset (i.e. not due to a degenerative disease such as ALS or MS) SCI (either traumatic or non-traumatic)
* Discharged from initial inpatient rehabilitation and living in the community for at least 3 months
* Age 18 or older at the time of enrollment
* Age at least 16 years at the time of their spinal cord injury
* Current symptoms (no more than two weeks from the time of consent) of at least mild depression and/or anxiety, as determined by a score of ≥5 on the eight-item Patient Health Questionnaire depression scale (PHQ-8) and/or seven-item Generalized Anxiety Disorder measure (GAD-7).

Exclusion Criteria:

* Male and female participants younger than 18 years old
* A lack of English proficiency needed to comprehend and complete study measures and review online study content.
* Current cognitive impairment that would limit comprehension of informed consent or study procedures, as determined by the member of the study team conducting informed consent.
* Lack of access to the internet and an internet-enabled computer or smart device.
* A spinal cord injury that is due to a degenerative disease (e.g. ALS, MS) and not sudden onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
Change in weekly depression symptoms as measured by the Spinal Cord Injury - Quality of Life (SCI-QOL) Depression computer adaptive test (CAT) | Weeks 1-6
  Patient-reported outcome measure of current depressive symptoms which is included in the intervention and control conditions each week.
Change in weekly anxiety symptoms as measured by the Spinal Cord Injury - Quality of Life (SCI-QOL) Anxiety computer adaptive test (CAT) | Weeks 1-6
  Patient-reported outcome measure of current anxiety symptoms which is included in the intervention and control conditions each week.

SECONDARY OUTCOMES:
Change in Current Depressive Symptoms as assessed by the Patient Health Questionnaire (PHQ)-8 | Change from Baseline to Week 6. Also used for screening.
  Patient-reported measure of depression
Change in Current Symptoms of anxiety as assessed by the Generalized Anxiety Disorder (GAD-7) | Change from Baseline to Week 6. Also used for screening.
  Patient-reported measure of depression
Change in weekly resilience levels as measured by the Spinal Cord Injury - Quality of Life (SCI-QOL) resilience computer adaptive test (CAT) | Weeks 1-6
  Patient-reported outcome measure of current resilience which is included in the intervention and control conditions each week.

OTHER OUTCOMES:
Qualitative information on the usability of the system as measured by a System Usability Survey | At the end of the final (6th) system session. Each system session is open for 4 days or until the participant completes the session, whichever comes first.
  Participants will complete a usability survey following the final session to provide information on the usability of the system.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware College of Health Sciences, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No